CLINICAL TRIAL: NCT00006049
Title: A Randomized, Double-Blind, Phase III Comparative Trial of 2 Doses of ZD1839 (IRESSA) in Combination With Paclitaxel and Carboplatin Versus Placebo in Combination With Paclitaxel and Carboplatin in Chemotherapy-Naive Patients With Advanced (Stage III or IV) Non-Small Cell Lung Cancer
Brief Title: ZD 1839 Plus Chemotherapy in Treating Patients With Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: AstraZeneca (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068065; ZENECA-1839IL/0017; MSKCC-00100
Record Dates: First submitted 2000-07-05; First posted 2004-04-26 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2001-07

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Gefitinib; Paclitaxel

INTERVENTIONS:
Drug: carboplatin
Drug: gefitinib
Drug: paclitaxel

SUMMARY:
RATIONALE: Some tumors need growth factors produced by the body's white blood cells to keep growing. ZD 1839 may interfere with the growth factor and stop the tumor from growing. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether combination chemotherapy is more effective with or without ZD 1839 for non-small cell lung cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of combination chemotherapy with or without ZD 1839 in treating patients who have stage III or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the 1 year survival rate, time to worsening of disease related symptoms, and progression free survival in chemotherapy naive patients with stage IIIB or IV non-small cell lung cancer treated with one of two doses of ZD 1839 or placebo combined with paclitaxel and carboplatin. II. Compare the quality of life of patients treated with these three regimens.

OUTLINE: This is a randomized, double blind, placebo controlled, multicenter study. Patients are randomized to one of three treatment arms. All patients receive paclitaxel IV over 3 hours followed by carboplatin IV over 15-30 minutes on day 1. Patients receive lower dose oral ZD 1839 (arm I), higher dose oral ZD 1839 (arm II), or placebo (arm III) twice on day 1, and then once daily thereafter. Chemotherapy repeats every 3 weeks for a maximum of 6 courses. ZD 1839 or placebo continues daily in the absence of disease progression or unacceptable toxicity. Quality of life is assessed prior to study, then every 3 weeks until completion of chemotherapy, then every 4 weeks until completion of oral ZD 1839 or placebo, and then every 8 weeks thereafter. Patients are followed every 8 weeks.

PROJECTED ACCRUAL: A total of 1,029 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven non-small cell lung cancer Stage III disease that is not curable with surgery or radiotherapy OR Stage IV disease Chemotherapy naive

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 2,000/mm3 WBC at least 4,000/mm3 Platelet count at least 100,000/mm3 Hepatic: ALT or AST no greater than 2.5 times upper limit of normal (ULN) (no greater than 5 times ULN if liver metastasis present) Renal: Creatinine no greater than 1.5 times ULN Cardiovascular: No evidence of severe or uncontrolled cardiovascular disease Pulmonary: No evidence of severe or uncontrolled pulmonary disease Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Endocrine therapy: No concurrent therapy that may interfere with evaluation of response Radiotherapy: See Disease Characteristics Prior localized irradiation allowed Surgery: See Disease Characteristics Prior surgery allowed Other: No concurrent drugs with known significant cytochrome P450 3A4 inhibitory effects (e.g., ketoconazole, itraconazole, troleandomycin, erythromycin, diltiazem, verapamil) No concurrent use of contact lenses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-05

CONTACTS AND LOCATIONS:
Overall Officials: Ron Staugarrd, Study Chair — AstraZeneca
Locations (1):
- AstraZeneca Pharmaceuticals LP, Wilmington, Delaware, United States